CLINICAL TRIAL: NCT04298996
Title: Effect of Passive Smoking on Oxidative Stress and Dental Caries in Children
Status: Completed | Type: Observational
Sponsor: Merve Erkmen Almaz (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Sponsor-Investigator, Merve Erkmen Almaz, Assist prof, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: 2016-140
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Oxidative Stress; Dental Caries; Passive Smoking
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group (passive smoking children): examining for caries prevalence and taking saliva samples to determine oxidative stress markers TAS and TOS
  Interventions: Diagnostic Test: taking saliva samples to determine oxidative stress markers TAS and TOS
- control group: examining for caries prevalence and taking saliva samples to determine oxidative stress markers TAS and TOS
  Interventions: Diagnostic Test: taking saliva samples to determine oxidative stress markers TAS and TOS

INTERVENTIONS:
Diagnostic Test: taking saliva samples to determine oxidative stress markers TAS and TOS

SUMMARY:
The purpose of the present study was to determine the effect of passive smoking on oxidative stress and dental caries in children.A total of 180 children were included to the study as follows; 90 children exposed to passive smoking, and 90 children in the control group (unexposed controls). Also demographic data were recorded (age, gender, parental education levels, child's tooth-brushing habit and child's daily dietary sugar exposure, family income). Dental examination of children were performed and caries prevalence of the patients were recorded. Unstimulated saliva samples were collected from children. Saliva 'cotinine levels' and oxidative stress markers 'total antioxidant status' (TAS), and' total oxidant status' (TOS) were evaluated by using Enzyme-linked immunosorbent assay (ELISA). The obtained data parameters of the two groups were evaluated and comparison was performed.

ELIGIBILITY:
Inclusion Criteria:

-Systemically healthy children

Exclusion Criteria:

* Uncooperative children
* The presence of orthodontic/intraoral appliance
* Any disease or condition known to affect oxidative stress

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children, referring for dental examination to the Department of Pediatric Dentistry of Kirikkale University, were selected.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
determining oxidative stress marker in saliva: TAS | 1 day (once after the dental examination)]
  Unstimulated saliva samples were collected from children.
determining oxidative stress marker in saliva: TOS | 1 day (once after the dental examination)
  Unstimulated saliva samples were collected from children.
determining caries prevalence | 1 day (once for dental examination)
  Children were examined to determine caries prevalence.